CLINICAL TRIAL: NCT07057752
Title: Effect of Virtual Reality Distraction in Reducing Patients' Pain and Anxiety During Peripheral Arterial Angioplasty: a Randomized Prospective Study
Brief Title: Virtual Reality for Pain and Anxiety Relief During Peripheral Angioplasty
Acronym: VRPAIN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, İsmail DAL, Assistant Professor Literally: Doctor Teaching Member, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KastamonuUni
Record Dates: First submitted 2025-06-22; First posted 2025-07-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Angioplasty; Pain Management; Virtual Reality
MeSH Terms: conditions — Agnosia | interventions — dexketoprofen trometamol; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Virtual reality glasses will be applied to patients in this group in addition to painkillers
  Interventions: Other: Virtual Reality
- Routine treatment group (Active Comparator): Patients in this group will be administered painkillers routinely in the hospital.
  Interventions: Drug: dexketoprofen + midazolam

INTERVENTIONS:
Other: Virtual Reality — Virtual reality (VR) will be applied to patients in this group in addition to painkillers. VR is a non-pharmacological method that uses special glasses to create an immersive visual and auditory experience. It helps distract patients from the procedure and may reduce pain and anxiety.
  Arms: Virtual Reality
Drug: dexketoprofen + midazolam — Patients in this group will be treated with dexketoprofen as a painkiller and midazolam as an anxiolytic, if needed. This combination aims to reduce both pain and anxiety during the procedure.
  Arms: Routine treatment group

SUMMARY:
Peripheral arterial disease can cause serious leg pain and discomfort. During treatment with angioplasty, patients often feel pain and anxiety because the procedure is usually done with local anesthesia and no sedation. Virtual reality (VR) may help reduce these feelings by distracting patients.

This study will test whether using VR glasses during peripheral angioplasty can lower patients' pain and anxiety. Patients will be randomly divided into two groups: one will use VR, the other will not. Pain and anxiety will be measured at different times during the procedure. The need for extra pain or anxiety medication and overall satisfaction will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective peripheral angioplasty
* Can cooperate and appropriate for wearing VR glasses

Exclusion Criteria:

* Undergoing emergency peripheral angioplasty
* With neurological and psychiatric conditions that prevent reliable assessment of pain or anxiety scores

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | 1 day
  Pain level will be measured with the Numerical Rating Scale (NRS). It ranges between minimum 0 and maximum 10 points. 0 point reffers no pain, 10 points reffer most serious pain.
State Anxiety Inventory-6 (STAI-6) | 1 day
  Anxiety level was measured with the State Anxiety Inventory-6 (STAI-6). After a correction formula it ranges between minimum 20 and maximum 80 points. 20 points reffer lower anxiety, 80 points reffer higher anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu Education and Research Hospital, Kastamonu, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
yes
Time Frame: Data will become available persistantly on 1.1.2026.
Access Criteria: Upon reasonable request principal investigator will share the data.